CLINICAL TRIAL: NCT06244368
Title: A Single Arm, Open Label, Multi-center Study of Mitoxantrone Hydrochloride Liposome, Gemcitabine, Vinorelbine With or Without Anti-CD20 Monoclonal Antibody (GVM±R) in Patients With Relapsed or Refractory Aggressive Non-Hodgkin's Lymphoma
Brief Title: GVM±R in Patients With Relapsed or Refractory Aggressive NHL.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: First Hospital of China Medical University (Other); Hebei Medical University Fourth Hospital (Other); Chengdu Shangjin Nanfu Hospital (Unknown); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Xuanwu Hospital, Beijing (Other); The Affiliated Ganzhou Hospital of Nanchang University (Other); Beijing Tongren Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); The First Hospital of Jilin University (Other); People's Hospital of Zhengzhou University (Other); The First Affiliated Hospital of Bengbu Medical University (Other); The Second Affiliated Hospital of Kunming Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Shengjing Hospital (Other); Peking University Third Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); China-Japan Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023065
Record Dates: First submitted 2024-01-28; First posted 2024-02-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Peripheral T Cell Lymphoma; Diffuse Large B-cell Lymphoma
Keywords: aggressive non-Hodgkin's lymphoma (NHL); Mitoxantrone hydrochloride liposome; GVM±R
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GVM±R (Experimental): Patients with relapsed or refractory aggressive NHL will undergo GVM±R therapy
  Interventions: Drug: GVM±R regimen

INTERVENTIONS:
Drug: GVM±R regimen — Mitoxantrone hydrochloride liposome (18 mg/m^2) on day 1； Gemcitabine (800 mg/m^2) on day 1,8； Vinorelbine (20mg/m^2) on day 1,8； Rituximab (375mg/m^2) on day 1;
  The regimen will be administered every 3 weeks, for a maximum of 6 cycles. The choice of CD20 monoclonal antibody will be determined by the attending physician.

SUMMARY:
This is a prospective clinical study to evaluate the safety and efficacy of GVM±R in patients with relapsed or refractory aggressive non-Hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
This is a single-arm, open label, multi-center clinical study to evaluate the safety and efficacy of mitoxantrone hydrochloride liposome in combination with gemcitabine, vinorelbine and/or anti-CD20 monoclonal antibody(GVM ± R) in patients with relapsed or refractory aggressive non-Hodgkin lymphoma (NHL).Mitoxantrone hydrochloride liposome will be given on day 1 at dose of 18 mg/m2 and be combined with gemcitabine, vinorelbine and/or rituximab (Pts with CD20-positive lymphomas are evaluated by the investigator on whether to combine rituximab or choose another CD20 monoclonal antibody).Each cycle consists of 21 days. A maximum of 6 cycles of therapy are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, ≤65 years.
2. Expected survival ≥ 3 months.
3. Subjects with aggressive NHL who have relapsed or proven refractory to at least one line of standard therapy or have achieved PR as the best response after a minimum of 4 cycles of therapy (patients with a Deauville score of 4 must have biopsy-proven residual disease). Relapse is defined as a disease response (PR/CR) to the last-line therapy with a duration of response exceeding 6 months. Refractory disease can be confirmed under any of the following conditions: 1) no partial or complete response to the last-line therapy; 2) the duration of complete or partial response to the last-line therapy is no longer than 6 months from the last dose of therapy; 3) Recurrence after hematopoietic stem cell transplantation.
4. Subjects must have at least one measurable lesion per lugano2014 criteria: for lymph node lesions, the long diameter should be > 1.5cm; For non-lymph node lesions, the long diameter should be > 1.0cm;
5. Eastern Cooperative Oncology Group (ECOG) : 0-2
6. Peripheral blood: Absolute neutrophil count (ANC) ≥1.5×109/L, Platelet count (PLT) ≥75×109/L, Hemoglobin(HB)≥ 80g/L.(Restriction may be relaxed in patients with bone marrow involvement, Absolute neutrophil count (ANC) ≥1.0×109/L, Platelet count (PLT) ≥50×109/L, Hemoglobin(HB)≥ 75g/L).
7. Liver and kidney function: Serum creatinine (Scr) ≤1.5X upper limit of normal (ULN).Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5X ULN, Total bilirubin (TBIL) ≤1.5X upper limit of normal (ULN).(If the lymphoma involves the liver, TBIL≤3 X ULN.AST and ALT≤5 X ULN). For Pts diagnosed with Gilbert's disease, TBIL was enrolled if it was ≤3 X ULN.-

Exclusion Criteria:

1. The subject had previously received any of the following anti-tumor treatments:

   1. Subjects who have been treated with mitoxantrone or mitoxantrone liposomes;
   2. Previously received doxorubicin or other anthracycline treatment, and the total cumulative dose of doxorubicin was more than 360 mg/m2 (For other anthracyclines, 1 mg doxorubicin equivalent to 2 mg epirubicin);
   3. Subjects who received anti-tumor treatment (including chemotherapy, targeted therapy, glucocorticoid, traditional Chinese medicine with anti-tumor activity, etc.) or participated in other clinical trials and received trial drugs within 4 weeks or 5 half-lives((whichever comes first) before the first administration of the study drugs;
   4. Subjects who received autologous hematopoietic stem cell transplantation or allogeneic hematopoietic stem cell transplantation within 100 days before the first administration of study drugs;
   5. Subjects who received chimeric antigen receptor T-cell (CAR-T) therapy.
2. Hypersensitivity to any study drug or its components.
3. Uncontrolled systemic diseases (such as active infection, uncontrolled hypertension, diabetes, etc.)
4. Heart function and disease meet one of the following conditions:

   1. Long QTc syndrome or QTc interval > 480 ms;
   2. Complete left bundle branch block, grade II or III atrioventricular block;
   3. Serious and uncontrolled arrhythmias requiring drug treatment;
   4. New York Heart Association grade ≥ III;
   5. Left Ventricular Ejection Fractions (LVEF)< 50%;
   6. A history of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities within 6 months before recruitment.
5. Active hepatitis B and C infection (defined as hepatitis B virus surface antigen positive and hepatitis B virus DNA higher than the Upper limit of normal(ULN); Hepatitis C virus antibody positive and hepatitis C virus RNA higher than the Upper limit of normal).
6. Human immunodeficiency virus (HIV) infection (defined as HIV antibody positive).
7. Patients with other malignant tumors, except for effectively controlled non-melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ or other tumors without treatment during the past 5 years.
8. Pregnant and lactating women and patients of childbearing age who are unwilling to take contraceptive measures.
9. ≥ Grade 3 neuritis.
10. Active central nervous system (CNS) lymphoma;
11. Unsuitable subjects for this study determined by the investigator. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to 2 years
  Response is assessed according to the lugano criteria

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | up to 2 years
  Response is assessed according to the lugano criteria
Progression-Free-Survival (PFS) | up to 2 years
  From the date of the first dose of therapy is given until disease progression, death or last follow-up
Overall survival (OS) | up to 2 years
  From the date of inclusion to date of death, irrespective of cause
Incidence of Treatment-Emergent Adverse Events | up to 2 years
  The adverse events were evaluated by NCI-CTCAE 5.0 standard Hematologic and non-hematologic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Wei Liu, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, CAMS & PUMC; Xiaojing Yan, Principal Investigator — First Hospital of China Medical University; HaiSheng、Chen Liu 、Huang, Principal Investigator — Hebei Medical University Fourth Hospital; Yongqian Jia, Principal Investigator — Chengdu Shangjin Nanfu Hospital; Yunhong Huang, Principal Investigator — Affiliated Cancer Hospital & Institute of Guizhou Medical University; Xiaobo Wang, Principal Investigator — The Second Affiliated Hospital of Dalian Medical University; Wanling Sun, Principal Investigator — Xuanwu Hospital, Beijing; Mingxing Zhong, Principal Investigator — The Affiliated Ganzhou Hospital of Nanchang University; Liang Wang, Principal Investigator — Beijing Tongren Hospital; Xiuli Sun, Principal Investigator — The First Affiliated Hospital of Dalian Medical University; Ou Bai, Principal Investigator — The First Hospital of Jilin University; Shuxia Guo, Principal Investigator — People's Hospital of Zhengzhou University; Yanli Yang, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University; Zeping Zhou, Principal Investigator — The Second Affiliated Hospital of Kunming Medical University; Fei Li, Principal Investigator — The First Affiliated Hospital of Nanchang University; Aichun Liu, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University; Aijun Liao, Principal Investigator — Shengjing Hospital; Hongmei Jing, Principal Investigator — Peking University Third Hospital; Shuye Wang, Principal Investigator — First Affiliated Hospital of Harbin Medical University; Zhenling Li, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, CAMS & PUMC, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No